CLINICAL TRIAL: NCT02076178
Title: A Phase IIa Study to Evaluate the Safety, Tolerability and Acceptability of Long Acting Injections of the HIV Integrase Inhibitor, GSK1265744, in HIV Uninfected Men (ECLAIR)
Brief Title: Study to Evaluate the Safety Tolerability and Acceptability of Long Acting Injections of the Human Immunodeficiency Virus (HIV) Integrase Inhibitor, GSK1265744, in HIV Uninfected Men (ECLAIR)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201120
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Results first posted 2017-12-15 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-10

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: Pre-Exposure Prophylaxis; HIV integrase; Intramuscular Injection; GSK1265744
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Participants will receive daily oral 744 (30 mg tablets) for 4 weeks, followed by a one week washout period followed by intra-muscular (IM) injections of 800 mg of 744 LA at three time points at 12 week intervals as: Week 5, Week 17, and Week 29
  Interventions: Drug: 744 Tablet; Drug: 744 LA Injection
- Arm 2 (Experimental): Participants will receive daily oral matching placebo for 4 weeks, followed by a one week washout period followed by intra-muscular (IM) injections of saline at three time points at 12 week intervals as: Week 5, Week 17, and Week 29
  Interventions: Drug: Placebo Tablet; Drug: Placebo Injection

INTERVENTIONS:
Drug: 744 Tablet — White to almost white oval shaped film coated 30 mg tablets for oral administration
  Arms: Arm 1
Drug: 744 LA Injection — Sterile white to slightly coloured suspension containing 200 mg/mL of 744 as free acid for administration by intramuscular (IM) injection
  Arms: Arm 1
Drug: Placebo Tablet — Microcrystalline cellulose, Opadry film-coating, white OY-S-28876
  Arms: Arm 2
Drug: Placebo Injection — Sterile saline 0.9% Sodium Chloride Injection
  Arms: Arm 2

SUMMARY:
This study is a Phase IIa, randomized, multi-site, two-arm, double-blinded study to evaluate the safety, tolerability, and acceptability of GSK1265744 long acting injectable formulation (744 LA) in adult male subjects. To evaluate the safety and tolerability of the injectable agent, 744 LA (800 milligrams (mg) dose administered at three time points at 12 week intervals) through Week 41 in HIV-uninfected men. Eligible participants will be randomized in a 5:1 ratio to receive 744 LA or matching placebo. Participants will receive daily oral 744 (30 mg tablets) or matching placebo for 4 weeks during the Oral Phase of the study, followed by a one week washout period. Following safety lab assessments from the Oral Phase, participants will enter the Injection Phase and receive Intramuscular (IM) injections of 744 LA or placebo at three time points at 12 week intervals. IM injections will consist of 800 mg of 744 or a matching control

ELIGIBILITY:
Inclusion Criteria:

* Non-reactive HIV test at screening or enrollment.
* Males 18 to 65 years old at the time of signing the informed consent.
* At risk of acquiring HIV, defined as having at least one casual sex partner in the past 24 months.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring at the time of screening.
* If participating in sexual activity with a female of child-bearing potential, men must agree to use condoms. Subjects who are sexual partners of females with child bearing potential must also agree to practice an acceptable method of contraception for the duration of the study, such as double barrier (male condom/spermicide, male condom/diaphragm) or female partner use of hormonal contraception, intrauterine device (IUD) or other method with published data showing that the lowest expected failure rate for that is less than 1% per year. All subjects participating in the study must be counseled on safer sexual practices including the use of effective barrier methods to minimize risk of HIV transmission.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Willing to undergo all required study procedures

Exclusion Criteria:

* One or more reactive HIV test results at screening or enrollment, even if HIV infection is not confirmed. Negative HIV Ribonucleic acid (RNA) must also be documented at screening.
* Assessed by the Investigator of Record or designee as being at "high risk" for HIV infection. This may include one or more of the following:

The negative partner in an HIV serodiscordant couple Men who exchange sex for goods or money Men who have engaged in unprotected receptive anal intercourse within the past 6 months Men who have had greater than 3 sexual partners within the past 3 months Men who have had a sexually transmitted disease within the past 6 months Any other behavior assessed by the investigator as "high risk"

* Co-enrollment in any other HIV interventional research study (provided by self-report or other available documentation) or prior enrollment and receipt of the active arm (i.e., NOT a placebo) of a HIV vaccine trial (provided by available documentation).
* Use of antiretroviral (ARV) therapy (e.g., for Post exposure prophylaxis (PEP) or Pre exposure prophylaxis (PrEP) in the past 30 days, five half-lives, or twice the duration of the biological effect of the applied treatment (whichever is longer) prior to study enrollment.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of drug or alcohol consumption that in the opinion of the Principal Investigator will interfere with study participation.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Any of the following laboratory values during the screening period. Positive Hepatitis C antibody result Positive Hepatitis B surface antigen (HBsAg) Hemoglobin less than 11 gram (g)/deci liter (dL) Absolute neutrophil count less than 750 cells/mm^3 Platelet count less than or equal to 100,000/mm^3 Presence of a coagulopathy as defined by an INR greater than 1.5 or a PTT greater than 45sec Calculated creatinine clearance less than 70 mL/minute using the Cockcroft-Gault equation A single repeat test is allowed during the Screening period to verify a result, with the exception of HIV tests.
* Subjects with an alanine aminotransferase (ALT), alkaline phosphatase (ALP) or bilirubin greater than or equal to1.5xULN (isolated bilirubin greater than 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35%).
* History of the following cardiac diseases: myocardial infarction, congestive heart failure, documented hypertrophic cardiomyopathy, sustained ventricular tachycardia.
* The subject's systolic blood pressure is outside the range of 90-160mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 45-100 beats per minute (bpm).
* Exclusion criteria for screening (ECG (a single repeat is allowed for eligibility determination) for Male Subjects:

Heart rate (A heart rate from 100 to 110 bpm can be rechecked within 30 minutes to verify eligibility)-less than 45 and greater than 100 bpm.

QRS duration-greater than 120 msec. QTc interval (B or F)-greater than 450 msec. Evidence of previous myocardial infarction (does not include ST segment changes associated with repolarization).

Any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher], Wolf Parkinson White [WPW] syndrome).

Sinus Pauses greater than 3 seconds. Any significant arrhythmia which, in the opinion of the principal investigator and medical monitor, will interfere with the safety for the individual subject.

Non-sustained or sustained ventricular tachycardia (greater than or equal to 3 consecutive ventricular ectopic beats).

* Ongoing intravenous drug use - episodic use or any use in the past 90 days is exclusionary (as assessed by the study investigator).
* The subject has a tattoo or other dermatological condition overlying the gluteus region which may interfere with interpretation of ISRs.
* Use of high dose aspirin or any other anticoagulant or antiplatelet medication that would interfere with the ability to receive intramuscular injections.
* Active skin disease or disorder (i.e., infection, inflammation, dermatitis, eczema, drug rash, psoriasis, urticaria). Mild cases of localized acne or folliculitis or other mild skin condition may not be exclusionary at the discretion of the Investigator of Record or Medical Monitor).

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2014-03-27 (Actual); Primary Completion 2015-05-15 (Actual); Study Completion 2016-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (8):
- United States (8):
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Santa Fe, New Mexico
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Newport News, Virginia

REFERENCES:
- [Derived] Murray MI, Markowitz M, Frank I, Grant RM, Mayer KH, Hudson KJ, Stancil BS, Ford SL, Patel P, Rinehart AR, Spreen WR, Margolis DA. Satisfaction and acceptability of cabotegravir long-acting injectable suspension for prevention of HIV: Patient perspectives from the ECLAIR trial. HIV Clin Trials. 2018 Aug;19(4):129-138. doi: 10.1080/15284336.2018.1511346. Epub 2018 Nov 16. PMID 30445896
- [Derived] Markowitz M, Frank I, Grant RM, Mayer KH, Elion R, Goldstein D, Fisher C, Sobieszczyk ME, Gallant JE, Van Tieu H, Weinberg W, Margolis DA, Hudson KJ, Stancil BS, Ford SL, Patel P, Gould E, Rinehart AR, Smith KY, Spreen WR. Safety and tolerability of long-acting cabotegravir injections in HIV-uninfected men (ECLAIR): a multicentre, double-blind, randomised, placebo-controlled, phase 2a trial. Lancet HIV. 2017 Aug;4(8):e331-e340. doi: 10.1016/S2352-3018(17)30068-1. Epub 2017 May 22. PMID 28546090

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 10 centers in United states. Participants who received study medication are being followed for 52 Weeks following their last injection while those in placebo group were followed until all participants completed Week 41. The first subject's first visit was 27-Mar-2014 and the last subject's last visit was 15-May-2015.
Pre-assignment Details: A total of 205 participants were screened of which 78 participants were not randomized. The remaining 127 participants were randomized to the study treatment who entered the oral and injection phase. Out of this, one participant randomized but withdrawn consent prior to treatment.
Groups:
- Placebo: Eligible participants received matching placebo tablets for 4 Week during the Oral Phase of the study, followed by a 1 Week washout period, to assess for safety and tolerability prior to receiving matching placebo injections [0.9 percent saline]. Following safety laboratory assessments from the Oral Phase, participants entered the Injection Phase and received intramuscular (IM) injection of placebo at 3 time points at 12 Week intervals (Week 5, Week 17, and Week 29). The IM injection consisted of 800 mg of placebo.
- Cabotegravir: Eligible participants received daily oral cabotegravir 30 milligrams (mg) tablets for 4 Week during the Oral Phase of the study, followed by a 1 Week washout period, to assess for safety and tolerability prior to receiving cabotegravir injections. Following safety laboratory assessments from the Oral Phase, participants entered the Injection Phase and received IM injections of cabotegravir or placebo at 3 time points at 12 Week intervals (Week 5, Week 17, and Week 29). The IM injections consisted of 800 mg of cabotegravir.
Period: Oral Phase
Arm/Group | Placebo | Cabotegravir
Started | 21 | 106
Completed | 21 | 94
Not Completed | 0 | 12
Not completed — Adverse Event | 0 | 7
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Physician Decision | 0 | 1
Period: Injection Phase
Arm/Group | Placebo | Cabotegravir
Started | 21 | 94
Completed | 20 | 87
Not Completed | 1 | 7
Not completed — Protocol defined stopping criteria | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Physician Decision | 0 | 3
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Eligible participants received matching placebo tablets for 4 Week during the Oral Phase of the study, followed by a 1 Week washout period, to assess for safety and tolerability prior to receiving matching placebo injections [0.9 percent saline]. Following safety laboratory assessments from the Oral Phase, participants entered the Injection Phase and received IM injection of placebo at 3 time points at 12 Week intervals (Week 5, Week 17, and Week 29). The IM injection consisted of 800 mg of placebo.
- Cabotegravir: Eligible participants received daily oral cabotegravir 30 mg tablets for 4 Week during the Oral Phase of the study, followed by a 1 Week washout period, to assess for safety and tolerability prior to receiving cabotegravir injections. Following safety laboratory assessments from the Oral Phase, participants entered the Injection Phase and received IM injections of cabotegravir or placebo at 3 time points at 12 Week intervals (Week 5, Week 17, and Week 29). The IM injections consisted of 800 mg of cabotegravir.
- Total: Total of all reporting groups
Arm/Group | Placebo | Cabotegravir | Total
Number analyzed (Participants) | 21 | 106 | 127
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: One participant randomized but withdrawn consent prior to treatment and not included in analysis for Age, continuous.
  Years
    number analyzed (Participants) | 21 | 105 | 126
    (all) | 33.7 (11.56) | 35.1 (11.75) | 34.9 (11.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 21 | 106 | 127
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 7 | 33 | 40
  American Indian or Alaska Native | 0 | 3 | 3
  Asian - Central/South Asian Heritage | 1 | 2 | 3
  Asian - East Asian Heritage | 1 | 2 | 3
  Asian - South East Asian Heritage | 0 | 1 | 1
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1
  White - Arabic/North African Heritage | 0 | 3 | 3
  White - White/Caucasian/European Heritage | 12 | 59 | 71
  Unknown | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Grade 2 or Higher Event in the Injection Phase
Description: Clinical adverse event (AE) were graded using the Division of Acquired Immunodeficiency Syndrome (DAIDS) table for grading the severity of adult and pediatric AE Version 1.0, December 2004; Clarification August 2009. The grades were: 1 (mild)=Symptoms causing no or minimal interference with usual social and functional activities; 2 (moderate)= Symptoms causing greater than minimal interference with usual social and functional activities; 3 (severe)= Symptoms causing inability to perform usual social and functional activities; 4 (potentially life threatening): Symptoms causing inability to perform basic self-care functions or medical or operative intervention indicated to prevent permanent impairment, persistent disability, or death. Data has been presented for any Grade 2 or higher event in the injection phase for injection phase (Week 5- Week 41).
Time Frame: Up to Week 41
Population: Safety Injection population was defined as all participants enrolled in the study who received at least one injection of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cabotegravir
Number analyzed (Participants) | 21 | 94
Participants | 10 | 75
Statistical Analysis 1: Comparison: Placebo vs Cabotegravir; Any Grade 2 or higher event, any Grade 2 or higher event Vs Cabotegravir; Test type: Superiority or Other; p < 0.01, Fisher Exact

2. Primary Outcome: Number of Participants Who Recieved Injection Site Reaction (ISR) Related Concomitant Medication in the Injection Phase
Description: The concurrent medications that were consumed by participants during the injection phase were of the class nervous system, musculo-skeletal system, genito urinary systems and sex hormones, various, respiratory system, dermatologicals, alimentary tract and metabolism, sensory organs, systemic hormonal preparations, excluding sex hormones, blood and blood forming organs, cardiovascular system. The participants who took medication from any of the above class of during the injection phase (Week 5-Week 41) have been presented.
Time Frame: Up to Week 41
Population: The randomized population was defined as all participants who met the study criteria and were randomly assigned to treatment in the study.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Eligible participants received matching placebo tablets for 4 Week during the Oral Phase of the study, followed by a 1 Week washout period, to assess for safety and tolerability prior to receiving matching placebo injections [0.9 percent saline]. Following safety laboratory assessments from the Oral Phase, participants entered the Injection Phase and received IM injection of placebo at 3 time points at 12W intervals (W5, W17, and W29). The IM injection consisted of 800 mg of placebo.
Arm/Group | Placebo | Cabotegravir
Number analyzed (Participants) | 21 | 106
Participants | 5 | 55

3. Primary Outcome: Number of Participants Who Experienced Grade 2 or Higher Laboratory Results in the Injection Phase
Description: The severity of laboratory results was graded according to the DAIDS table for grading the severity of adult and pediatric AE Version 1.0, December 2004; Clarification August 2009. The DAIDS displays events as Grades 1-5 based on this general guideline: Grade 1, mild; Grade 2, moderate; Grade 3, severe; Grade 4, potentially life threatening. Data for Number of participants who experienced grade 2 or higher laboratory results in the injection phase (Week 5-Week 14) have been presented.
Time Frame: Up to Week 41
Population: Safety Injection population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cabotegravir
Number analyzed (Participants) | 21 | 94
Participants
  Activated prothrombin time/standard | 1 | 0
  Activated partial thromboplastin time | 1 | 0
  Alanine aminotransferase | 0 | 2
  Aspartate aminotransferase | 0 | 2
  Bilirubin | 0 | 4
  Carbon dioxide | 0 | 1
  Cholesterol | 1 | 4
  Creatine kinase | 3 | 6
  Glucose | 2 | 7
  Leukocytes | 0 | 2
  Lipase | 1 | 10
  Neutrophils | 0 | 3
  Prothrombin time | 1 | 0
  Urate | 1 | 0

4. Primary Outcome: Number of Participants Who Had Abnormal Electrocardiogram (ECG) Findings in the Injection Phase
Description: Full 12-lead ECGs included heart rate, PR, QRS, QT and QTc intervals. Measurements were taken from the participant following 5 minutes of rest in a semi-supine position. ECGs were performed at Week 5, Week 17, Week 29 and Week 41 in the injection phase (Week 5-Week 41). ECG abnormalities characterized as abnormal-not clinically significant (A-NCS) and abnormal-clinically significant (A-CS) upto Week 41 have been presented. There were no A-CS findings for ECG in the injection phase.
Time Frame: Up to Week 41
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cabotegravir
Number analyzed (Participants) | 21 | 105
Participants
  Week 5, A-NCS: number analyzed (Participants) | 21 | 93
  Week 5, A-NCS | 6 | 30
  Week 17, A-NCS: number analyzed (Participants) | 21 | 91
  Week 17, A-NCS | 9 | 34
  Week 29, A-NCS: number analyzed (Participants) | 20 | 87
  Week 29, A-NCS | 7 | 27
  Week 41, A-NCS: number analyzed (Participants) | 20 | 91
  Week 41, A-NCS | 5 | 23

5. Primary Outcome: Change From Baseline in Vital Sign Assessment for Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) in the Injection Phase
Description: Vital signs measurements were performed for SBP and DBP following 5 minutes of rest. Baseline was defined as the first injection at Week 5 for the injection phase. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline value at Week 17, Week 29 and Week 41.
Time Frame: Baseline (Week 5) to Week 41
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Placebo | Cabotegravir
Number analyzed (Participants) | 21 | 105
millimeters of mercury
  Week 17, DBP: number analyzed (Participants) | 21 | 91
  Week 17, DBP | -3.10 (11.541) | -0.74 (7.214)
  Week 29, DBP: number analyzed (Participants) | 20 | 87
  Week 29, DBP | -3.75 (12.781) | 0.32 (8.283)
  Week 41, DBP: number analyzed (Participants) | 21 | 92
  Week 41, DBP | -1.19 (13.692) | 0.01 (9.286)
  Week 17, SBP: number analyzed (Participants) | 21 | 91
  Week 17, SBP | -1.52 (14.041) | -0.66 (9.237)
  Week 29, SBP: number analyzed (Participants) | 20 | 87
  Week 29, SBP | 2.80 (10.904) | 2.62 (10.868)
  Week 41, SBP,: number analyzed (Participants) | 21 | 92
  Week 41, SBP, | -1.38 (14.044) | 1.64 (12.012)

6. Primary Outcome: Change From Baseline in Vital Sign Assessment for Heart Rate (HR) in the Injection Phase
Description: Vital signs measurements were performed for HR following 5 minutes of rest. Baseline was defined as the first injection at Week 5 for the injection phase. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline value at Week 17, Week 29 and Week 41.
Time Frame: Baseline (Week 5) to Week 41
Population: Safety population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Cabotegravir
Number analyzed (Participants) | 21 | 105
beats per minute
  Week 17, HR: number analyzed (Participants) | 21 | 91
  Week 17, HR | 1.19 (11.021) | 3.26 (11.684)
  Week 29, HR: number analyzed (Participants) | 20 | 87
  Week 29, HR | 1.55 (10.149) | 4.06 (10.740)
  Week 41, HR: number analyzed (Participants) | 21 | 92
  Week 41, HR | 1.43 (10.181) | 2.73 (11.752)

7. Primary Outcome: Number of Participant With ISR for the Injection Phase Defined by Maximum Grades
Description: Common ISR included pain, erythema, nodules and any other ISR with greater or equal to 5 participants. The number of participants who experienced pain events by needle length, swelling events by needle length, bump events by needle length for injection phase by maximum grades have been presented for the injection phase (Week 5-Week 41).
Time Frame: Up to Week 41
Population: Safety Injection population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cabotegravir
Number analyzed (Participants) | 21 | 94
Participants
  ISR pain, Grade 1 | 11 | 31
  ISR pain, Grade 2 | 1 | 37
  ISR pain, Grade 3 | 0 | 18
  ISR pain, Grade 4 | 0 | 0
  ISR swelling, Grade 1 | 0 | 11
  ISR swelling, Grade 2 | 0 | 4
  ISR swelling, Grade 3 | 0 | 0
  ISR swelling, Grade 4 | 0 | 0
  ISR Bump, Grade 1 | 0 | 9
  ISR Bump, Grade 2 | 0 | 3
  ISR Bump, Grade 3 | 0 | 0
  ISR Bump, Grade 4 | 0 | 0

8. Secondary Outcome: Plasma Pharmacokinetic Assessment for Area Under the Plasma Concentration-time Curve Over the Dosing Interval [AUC(0-tau)] in the Injection Phase
Description: Blood samples for pharmacokinetic analysis were collected starting on the first day of the First Injection Phase prior to the injection. At each injection visit a blood sample was collected prior to the injection at Week 5, Week 17 and Week 29, 1 Week post-injection at Week 6, Week 18, and Week 30, and 12 Week post-injection at Week 17, Week 29, and Week 41. The sample collected 12 Week following each injection served as the pre-dose sample for the subsequent dosing interval. Two additional samples were collected 4 and 8 Week after the first injection (Week 9 and Week 13), and 1 additional sample was collected 6 Week following the second and third injections (Week 23 and Week 35). Assessment was carried out for AUC(0-tau) a measure of the amount of drug available at target tissue (in plasma) for a fixed dosing interval (i.e.12 hours).
Time Frame: Up to Week 41
Population: The pharmacokinetic parameter population comprised of all participants who underwent plasma pharmacokinetic sampling and have evaluable cabotegravir parameters estimated. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram per milliliter
Arm/Group | Cabotegravir
Number analyzed (Participants) | 93
hour*microgram per milliliter
  Injection 1 | 3414.71 (42.5)
  Injection 2: number analyzed (Participants) | 89
  Injection 2 | 3873.25 (44.3)
  Injection 3: number analyzed (Participants) | 85
  Injection 3 | 4020.89 (36.2)

9. Secondary Outcome: Plasma Pharmacokinetic Assessment for Concentration at the End of the Dosing Interval (Ctau) and Maximum Observed Concentration (Cmax) in the Injection Phase
Description: Blood samples for pharmacokinetic analysis were collected starting on the first day of the First Injection Phase prior to the injection. At each injection visit a blood sample was collected prior to the injection at Week 5, Week 17 and Week 29, 1 Week post-injection at Week 6, Week 18, and Week 30, and 12 Week post-injection at Week 17, Week 29, and Week 41. The sample collected 12 Week following each injection served as the pre-dose sample for the subsequent dosing interval. Two additional samples were collected 4 and 8 Week after the first injection (Week 9 and Week 13), and 1 additional sample was collected 6 Week following the second and third injections (Week 23 and Week 35). Assessment was carried out for Ctau defined as the concentration at the end of the dosing interval and Cmax defined as the maximum observed plasma concentration.
Time Frame: Up to Week 41
Population: Pharmacokinetic parameter population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter
Arm/Group | Cabotegravir
Number analyzed (Participants) | 94
micrograms per milliliter
  Cmax, Injection 1: number analyzed (Participants) | 93
  Cmax, Injection 1 | 4.26 (88.6)
  Cmax, Injection 2: number analyzed (Participants) | 89
  Cmax, Injection 2 | 5.22 (78.0)
  Cmax, Injection 3: number analyzed (Participants) | 85
  Cmax, Injection 3 | 4.91 (66.6)
  Ctau, Injection 1: number analyzed (Participants) | 84
  Ctau, Injection 1 | 0.302 (157.1)
  Ctau, Injection 2: number analyzed (Participants) | 71
  Ctau, Injection 2 | 0.331 (164.5)
  Ctau, Injection 3: number analyzed (Participants) | 66
  Ctau, Injection 3 | 0.387 (149.6)

10. Secondary Outcome: Plasma Pharmacokinetic Assessment for Time to Maximum Observed Concentration (Tmax), Apparent Terminal Phase Half-life for (t½) in the Injection Phase
Description: Blood samples for pharmacokinetic analysis were collected starting on the first day of the First Injection Phase prior to the injection. At each injection visit a blood sample was collected prior to the injection at Week 5, Week 17 and Week 29, 1 Week post-injection at Week 6, Week 18, and Week 30, and 12 Week post-injection at Week 17, Week 29, and Week 41. The sample collected 12 Week following each injection served as the pre-dose sample for the subsequent dosing interval. Two additional samples were collected 4 and 8 Week after the first injection (Week 9 and Week 13), and 1 additional sample was collected 6 Week following the second and third injections (Week 23 and Week 35). Assessment was carried out for tmax defined as the time to the maximum observed plasma concentration and t½ defined as the time taken for the concentration of drug in the blood to decrease by half of the original amount.
Time Frame: Up to Week 41
Population: Pharmacokinetic parameter population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Cabotegravir
Number analyzed (Participants) | 93
days
  tmax, Injection 1 | 13.14 (11.503)
  tmax, Injection 2: number analyzed (Participants) | 89
  tmax, Injection 2 | 8.91 (9.311)
  tmax, Injection 3: number analyzed (Participants) | 85
  tmax, Injection 3 | 9.25 (7.579)
  t½ , Injection 1: number analyzed (Participants) | 61
  t½ , Injection 1 | 20.54 (10.690)
  t½ , Injection 2: number analyzed (Participants) | 0
  t½ , Injection 3: number analyzed (Participants) | 0

11. Secondary Outcome: Plasma Pharmacokinetic Assessment for AUC(0-tau) by Demographic Factor Body Mass Index (BMI) and Needle Length in the Injection Phase
Description: The median BMI was 26 kilogram per meter square. Plasma pharmacokinetic assessments were performed for AUC (0-tau) by BMI, either above or below the median BMI (50 percent upper and lower, where upper summary included all participants with BMI greater than or equal to the median BMI of the population and lower summary included all participants with BMI below the median BMI). Assessments was also performed for AUC (0-tau) by needle length (1.5 inch and 2 inch). Needle length and BMI were correlated in that the longer needle was recommended for participants with BMI greater than 30 kilogram per meter square.
Time Frame: Up to Week 41
Population: Pharmacokinetic parameter population. Only those participants available at the specified time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram per milliter
Arm/Group | Cabotegravir
Number analyzed (Participants) | 93
hour*microgram per milliter
  50 percent BMI lower, Injection 1: number analyzed (Participants) | 47
  50 percent BMI lower, Injection 1 | 4103.71 (28.4)
  50 percent BMI lower, Injection 2: number analyzed (Participants) | 44
  50 percent BMI lower, Injection 2 | 4250.82 (49.6)
  50 percent BMI lower, Injection 3: number analyzed (Participants) | 40
  50 percent BMI lower, Injection 3 | 4847.07 (26.1)
  50 percent BMI upper, Injection 1: number analyzed (Participants) | 46
  50 percent BMI upper, Injection 1 | 2830.06 (45.6)
  50 percent BMI upper, Injection 2: number analyzed (Participants) | 45
  50 percent BMI upper, Injection 2 | 3536.52 (36.7)
  50 percent BMI upper, Injection 3: number analyzed (Participants) | 45
  50 percent BMI upper, Injection 3 | 3405.52 (35.2)
  1.5 inch Injection 1: number analyzed (Participants) | 69
  1.5 inch Injection 1 | 3666.95 (40.0)
  1.5 inch Injection 2: number analyzed (Participants) | 64
  1.5 inch Injection 2 | 4177.42 (44.0)
  1.5 inch Injection 3: number analyzed (Participants) | 60
  1.5 inch Injection 3 | 4263.31 (38.9)
  2 inch Injection 1: number analyzed (Participants) | 24
  2 inch Injection 1 | 2782.06 (42.6)
  2 inch Injection 2: number analyzed (Participants) | 25
  2 inch Injection 2 | 3191.72 (38.5)
  2 inch Injection 3: number analyzed (Participants) | 25
  2 inch Injection 3 | 3493.85 (24.1)

12. Secondary Outcome: Plasma Pharmacokinetic Assessment for Ctau and Cmax by Demographic Factor BMI and Needle Length in the Injection Phase
Description: The median BMI was 26 kilogram per meter square. Plasma pharmacokinetic assessments were performed for Ctau and Cmax by BMI, either above or below the median BMI (50 percent upper and lower, where upper summary included all participants with BMI greater than or equal to the median BMI of the population and lower summary included all participants with BMI below the median BMI.
  ). Assessments was also performed for Ctau and Cmax by needle length (1.5 inch and 2 inch). Needle length and BMI were correlated in that the longer needle was recommended for participants with BMI greater than 30 kilogram per meter square.
Time Frame: Up to Week 41
Population: Pharmacokinetic parameter population. Only those participants available at the specified time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliter
Arm/Group | Cabotegravir
Number analyzed (Participants) | 93
micrograms per milliter
  50 percent BMI lower for Cmax, Injection 1: number analyzed (Participants) | 47
  50 percent BMI lower for Cmax, Injection 1 | 6.02 (51.3)
  50 percent BMI lower for Cmax, Injection 2: number analyzed (Participants) | 44
  50 percent BMI lower for Cmax, Injection 2 | 6.65 (54.8)
  50 percent BMI lower for Cmax, Injection 3: number analyzed (Participants) | 40
  50 percent BMI lower for Cmax, Injection 3 | 6.99 (35.9)
  50 percent BMI lower for Ctau, Injection 1: number analyzed (Participants) | 40
  50 percent BMI lower for Ctau, Injection 1 | 0.226 (159.9)
  50 percent BMI lower for Ctau, Injection 2: number analyzed (Participants) | 34
  50 percent BMI lower for Ctau, Injection 2 | 0.312 (138.3)
  50 percent BMI lower for Ctau, Injection 3: number analyzed (Participants) | 30
  50 percent BMI lower for Ctau, Injection 3 | 0.334 (102.2)
  50 percent BMI upper for Cmax, Injection 1: number analyzed (Participants) | 46
  50 percent BMI upper for Cmax, Injection 1 | 2.99 (100.0)
  50 percent BMI upper for Cmax, Injection 2: number analyzed (Participants) | 45
  50 percent BMI upper for Cmax, Injection 2 | 4.12 (88.4)
  50 percent BMI upper for Cmax, Injection 3: number analyzed (Participants) | 45
  50 percent BMI upper for Cmax, Injection 3 | 3.59 (68.0)
  50 percent BMI upper for Ctau, Injection 1: number analyzed (Participants) | 44
  50 percent BMI upper for Ctau, Injection 1 | 0.394 (141.7)
  50 percent BMI upper for Ctau, Injection 2: number analyzed (Participants) | 37
  50 percent BMI upper for Ctau, Injection 2 | 0.350 (193.8)
  50 percent BMI upper for Ctau, Injection 3: number analyzed (Participants) | 36
  50 percent BMI upper for Ctau, Injection 3 | 0.437 (193.3)
  1.5 inch for Cmax, Injection 1: number analyzed (Participants) | 69
  1.5 inch for Cmax, Injection 1 | 4.94 (79.3)
  1.5 inch for Cmax, Injection 2: number analyzed (Participants) | 64
  1.5 inch for Cmax, Injection 2 | 6.09 (63.7)
  1.5 inch for Cmax, Injection 3: number analyzed (Participants) | 60
  1.5 inch for Cmax, Injection 3 | 5.56 (65.0)
  1.5 inch for Ctau, Injection 1: number analyzed (Participants) | 62
  1.5 inch for Ctau, Injection 1 | 0.270 (177.7)
  1.5 inch for Ctau, Injection 2: number analyzed (Participants) | 50
  1.5 inch for Ctau, Injection 2 | 0.312 (152.4)
  1.5 inch for Ctau, Injection 3: number analyzed (Participants) | 47
  1.5 inch for Ctau, Injection 3 | 0.372 (150.7)
  2 inch for Cmax, Injection 1: number analyzed (Participants) | 24
  2 inch for Cmax, Injection 1 | 2.78 (92.8)
  2 inch for Cmax, Injection 2: number analyzed (Participants) | 25
  2 inch for Cmax, Injection 2 | 3.52 (92.7)
  2 inch for Cmax, Injection 3: number analyzed (Participants) | 25
  2 inch for Cmax, Injection 3 | 3.65 (57.6)
  2 inch for Ctau, Injection 1: number analyzed (Participants) | 22
  2 inch for Ctau, Injection 1 | 0.418 (93.7)
  2 inch for Ctau, Injection 2: number analyzed (Participants) | 21
  2 inch for Ctau, Injection 2 | 0.381 (200.3)
  2 inch for Ctau, Injection 3: number analyzed (Participants) | 19
  2 inch for Ctau, Injection 3 | 0.426 (152.1)

13. Secondary Outcome: Plasma Pharmacokinetic Assessment for Tmax and t½ by Demographic Factor BMI and Needle Length in the Injection Phase
Description: The median BMI was 26 kilogram per meter square. Plasma pharmacokinetic assessments were performed for tmax and t½ by BMI, either above or below the median BMI (50 percent upper and lower, where upper summary included all participants with BMI greater than or equal to the median BMI of the population and lower summary included all participants with BMI below the median BMI). Assessments was also performed for tmax and t½ by needle length (1.5 inch and 2 inch). Needle length and BMI were correlated in that the longer needle was recommended for participants with BMI greater than 30 kilogram per meter square.
Time Frame: Up to Week 41
Population: Pharmacokinetic parameter population. Only those participants available at the specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cabotegravir
Number analyzed (Participants) | 93
Days
  50 percent BMI lower for tmax, Injection 1: number analyzed (Participants) | 47
  50 percent BMI lower for tmax, Injection 1 | 8.55 (5.402)
  50 percent BMI lower for tmax, Injection 2: number analyzed (Participants) | 44
  50 percent BMI lower for tmax, Injection 2 | 8.62 (7.378)
  50 percent BMI lower for tmax, Injection 3: number analyzed (Participants) | 40
  50 percent BMI lower for tmax, Injection 3 | 7.75 (1.845)
  50 percent BMI lower for t½, Injection 1: number analyzed (Participants) | 39
  50 percent BMI lower for t½, Injection 1 | 19.54 (10.384)
  50 percent BMI lower for t½, Injection 2: number analyzed (Participants) | 0
  50 percent BMI lower for t½, Injection 3: number analyzed (Participants) | 0
  50 percent BMI upper for tmax, Injection 1: number analyzed (Participants) | 46
  50 percent BMI upper for tmax, Injection 1 | 17.83 (14.008)
  50 percent BMI upper for tmax, Injection 2: number analyzed (Participants) | 45
  50 percent BMI upper for tmax, Injection 2 | 9.20 (10.955)
  50 percent BMI upper for tmax, Injection 3: number analyzed (Participants) | 45
  50 percent BMI upper for tmax, Injection 3 | 10.58 (10.139)
  50 percent BMI upper for t½, Injection 1: number analyzed (Participants) | 22
  50 percent BMI upper for t½, Injection 1 | 22.32 (11.234)
  50 percent BMI upper for t½, Injection 2: number analyzed (Participants) | 0
  50 percent BMI upper for t½, Injection 3: number analyzed (Participants) | 0
  1.5 inch for tmax, Injection 1: number analyzed (Participants) | 69
  1.5 inch for tmax, Injection 1 | 11.33 (9.497)
  1.5 inch for tmax, Injection 2: number analyzed (Participants) | 64
  1.5 inch for tmax, Injection 2 | 9.10 (10.408)
  1.5 inch for tmax, Injection 3: number analyzed (Participants) | 60
  1.5 inch for tmax, Injection 3 | 9.53 (7.774)
  1.5 inch for t½, Injection 1: number analyzed (Participants) | 50
  1.5 inch for t½, Injection 1 | 21.26 (11.506)
  1.5 inch for t½, Injection 2: number analyzed (Participants) | 0
  1.5 inch for t½, Injection 3: number analyzed (Participants) | 0
  2 inch for tmax, Injection 1: number analyzed (Participants) | 24
  2 inch for tmax, Injection 1 | 18.34 (14.987)
  2 inch for tmax, Injection 2: number analyzed (Participants) | 25
  2 inch for tmax, Injection 2 | 8.42 (5.757)
  2 inch for tmax, Injection 3: number analyzed (Participants) | 25
  2 inch for tmax, Injection 3 | 8.57 (7.196)
  2 inch for t½, Injection 1: number analyzed (Participants) | 11
  2 inch for t½, Injection 1 | 17.27 (4.747)
  2 inch for t½, Injection 2: number analyzed (Participants) | 0
  2 inch for t½, Injection 3: number analyzed (Participants) | 0

14. Secondary Outcome: Number of Participants With Severity of ISRs and ISR Symptoms for Injection Phase Defined by Grades and Needle Length
Description: Acceptability of cabetogravir injections was assessed number of participants who had severe ISRs and ISR symptom. ISR examination for severity included an assessment of pain, pruritis, warm to touch, bruising, discoloration, erythema, swelling, induration and bump events. Common ISR Symptoms for Injection Phase included pain, erythema, nodules and any other ISRs with greater or equal to five participants. Data has been presented for the injection phase (W5-W41) by grades and needle length.
Time Frame: Up to Week 41
Population: Safety injection population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cabotegravir
Number analyzed (Participants) | 21 | 94
Participants
  ISR, needle any length, Pain, Grade 1, | 11 | 63
  ISR, needle any length, Pain, Grade 2 | 1 | 51
  ISR, needle any length, Pain, Grade 3 | 0 | 18
  ISR, needle any length, Pain, Grade 4 | 0 | 0
  ISR, needle any length, Pruritis, Grade 1 | 3 | 15
  ISR, needle any length, Pruritis, Grade 2 | 0 | 6
  ISR, needle any length, Pruritis, Grade 3 | 0 | 0
  ISR, needle any length, Pruritis, Grade 4 | 0 | 0
  ISR, needle any length, Bruising | 1 | 11
  ISR, needle any length, Discolouration | 0 | 4
  ISR, needle any length, Erythema | 0 | 6
  ISR, needle any length, Haemorrhage | 1 | 0
  ISR, needle any length, Induration | 0 | 10
  ISR, needle any length, Swelling | 0 | 15
  ISR, needle any length, Bump | 0 | 12
  ISR, needle any length, Warm to touch | 0 | 12
  ISR symptoms, needle any length, Mild or Grade 1 | 11 | 12
  ISR symptoms,needle any length,Moderate or Grade2 | 1 | 8
  ISR symptoms, needle any length, Severe or Grade 3 | 0 | 2
  ISR symptoms, needle any length, Grade 4 | 0 | 0

15. Secondary Outcome: Number of Participants With AE, Grade 2-4 AE and Serious Adverse Events (SAE) in the Oral Phase
Description: Clinical AE were graded using the DAIDS table for grading the severity of adult and pediatric AE Version 1.0, December 2004; Clarification August 2009. The grades were: 1 (mild)=Symptoms causing no or minimal interference with usual social and functional activities; 2 (moderate)= Symptoms causing greater than minimal interference with usual social and functional activities; 3 (severe)= Symptoms causing inability to perform usual social and functional activities; 4 (potentially life threatening): Symptoms causing inability to perform basic self-care functions or medical or operative intervention indicated to prevent permanent impairment, persistent disability, or death. Data has been presented for any Grade 2 or higher event in the injection phase for injection phase (Week 5- Week 41).
Time Frame: Up to Week 4
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cabotegravir
Number analyzed (Participants) | 21 | 105
Participants
  Any AE | 8 | 56
  Grade 2-4 AE | 4 | 24
  Any SAE | 0 | 0

16. Secondary Outcome: Number of Participants Who Received Concurrent Medication in Overall Study Duration
Description: The concurrent medications that were consumed by participants during the injection phase were of the class nervous system, musculo-skeletal system, genito-urinary systems and sex hormones, various, respiratory system, dermatologicals, alimentary tract and metabolism, anti-infectives for systemic use, sensory organs, systemic hormonal preparations excluding sex hormones, blood and blood forming organs, cardiovascular system, anti-neoplastic and immunomodulating agents, anti-parasitic products, insecticides and repellents . The participants who took medication from any of the above class of during the during the overall study duration injection phase (Day 1 until Week 41) have been presented.
Time Frame: Up to Week 41
Population: The Randomized Population comprised of all participants who met study criteria were randomly assigned to treatment in the study with the exception of any participants with documented evidence of not having consumed any amount of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cabotegravir
Number analyzed (Participants) | 21 | 106
Participants | 20 | 97

17. Secondary Outcome: Number of Participants Who Experienced Maximum Clinical Chemistry Including Liver Chemistry and Hematology Toxicities in the Oral Phase by Grades
Description: The severity of clinical chemistry including liver chemistry and hematology toxicities was graded according to the DAIDS table for grading the severity of adult and pediatric AE Version 1.0, December 2004; Clarification August 2009. The DAIDS displays events as Grades 1-5 based on this general guideline: Grade 1, mild; Grade 2, moderate; Grade 3, severe; Grade 4, potentially life threatening. Data for maximum clinical chemistry and hematology toxicities for oral phase (Day 1 upto Week 4) by grades have been presented.
Time Frame: Up to Week 4
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Cabotegravir
Number analyzed (Participants) | 21 | 105
Participants
  Clinical chemistry, Grade 1 | 2 | 33
  Clinical chemistry, Grade 2 | 3 | 4
  Clinical chemistry, Grade 3 | 0 | 2
  Clinical chemistry, Grade 4 | 0 | 4
  Liver chemistry, Grade 1 | 0 | 9
  Liver chemistry, Grade 2 | 0 | 2
  Liver chemistry, Grade 3 | 0 | 0
  Liver chemistry, Grade 4 | 0 | 1
  Hematology, Grade 1 | 0 | 4
  Hematology, Grade 3 | 0 | 0
  Hematology, Grade 2 | 0 | 1
  Hematology, Grade 4 | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to Week 41
Description: The safety population was used for analysis.
Arm/Group | Placebo | Cabotegravir
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/105
Serious Adverse Events (participants affected / at risk) | 1/21 | 1/105
Other Adverse Events (participants affected / at risk) | 18/21 | 100/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=21) | Cabotegravir (N=105)
Appendicitis (Infections and infestations) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=21) | Cabotegravir (N=105)
Injection site pain (General disorders) | 12 | 86
Injection site pruritus (General disorders) | 3 | 18
Injection site swelling (General disorders) | 0 | 20
Pyrexia (General disorders) | 1 | 17
Fatigue (General disorders) | 1 | 16
Injection site bruising (General disorders) | 1 | 11
Injection site warmth (General disorders) | 0 | 12
Injection site induration (General disorders) | 0 | 10
Chills (General disorders) | 0 | 6
Injection site erythema (General disorders) | 0 | 6
Upper respiratory tract infection (Infections and infestations) | 6 | 20
Nasopharyngitis (Infections and infestations) | 1 | 13
Viral upper respiratory tract infection (Infections and infestations) | 1 | 11
Gastroenteritis (Infections and infestations) | 0 | 6
Sinusitis (Infections and infestations) | 2 | 1
Headache (Nervous system disorders) | 4 | 26
Dizziness (Nervous system disorders) | 0 | 6
Diarrhoea (Gastrointestinal disorders) | 3 | 16
Nausea (Gastrointestinal disorders) | 2 | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 10
Blood creatine phosphokinase increased (Investigations) | 2 | 8
Neutropenia (Blood and lymphatic system disorders) | 0 | 8
Seasonal allergy (Immune system disorders) | 1 | 7
Insomnia (Psychiatric disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
The results are presented till Week 41 with cutoff date 15-May-2015.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.